CLINICAL TRIAL: NCT01940159
Title: A Randomized Single-Blind, Placebo-Controlled, Ascending Single Oral Dose Study Assessing the Safety, Tolerability, and Pharmacokinetics of SEP-363856 in Male and Female Subjects With Schizophrenia.
Brief Title: A Study Assessing the Safety, Tolerability, and Pharmacokinetics of SEP-363856 in Male and Female Subjects With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SEP361-105
Record Dates: First submitted 2013-09-06; First posted 2013-09-12 (Estimated); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Schizoaffective disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — SEP-363856

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Comparator: SEP-363856 (Active Comparator): Dosing will be initiated at 25 mg SEP-363856 as a single oral dose. Subsequent cohorts will be dosed at 50, 100, and 150 mg of SEP-363856
  Interventions: Drug: SEP-363856
- Placebo (Placebo Comparator): Matched placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SEP-363856 — SEP-36385625 as a single oral dose of 25, 50, 100, and 150 mcg
  Arms: Active Comparator: SEP-363856
Drug: Placebo — single oral dose placebo
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, single-blind, placebo-controlled, ascending single oral dose study designed to evaluate the safety, tolerability, and pharmacokinetic (PK) profiles of SEP-363856 and its metabolite SEP-363854 in male and female subjects with schizophrenia.

DETAILED DESCRIPTION:
This is a single-center, randomized, single-blind, placebo-controlled, ascending single oral dose study designed to evaluate the safety, tolerability, and PK of SEP-363856 and its metabolite SEP-363854 in male and female subjects with schizophrenia. This study will determine the maximum-tolerated dose (MTD) for a single oral dose of SEP-363856, and characterize the plasma PK profiles of SEP-363856 and its metabolite SEP-363854 in male and female subjects with schizophrenia.

For each of the dose-escalation cohorts, 12 subjects (9 active subjects and 3 placebo subjects) will receive a single oral dose. An attempt will be made to have at least one-third of subjects in each cohort be female.

Each cohort will be comprised of 12 subjects (9 active, 3 placebo). Within each cohort, subjects will be randomized to receive either SEP-363856 (active) or matched placebo in a 3:1 ratio.

The planned dose levels that will be evaluated are:

* Cohort 1: A single oral 25 mg dose of SEP-363856 or matched placebo.
* Cohort 2: A single oral 50 mg dose of SEP-363856 or matched placebo.
* Cohort 3: A single oral 100 mg dose of SEP-363856 or matched placebo.
* Cohort 4: A single oral 150 mg dose of SEP-363856 or matched placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must give written informed consent and privacy authorization (Healthcare Insurance, Portability, and Accountability Act of 1996) prior to participation in the study. Female subjects of childbearing potential and male subjects must agree to contraceptive requirements outlined in the informed consent form.
2. Subject must be willing and able to comply with the study procedures and visit schedules and must be able to follow verbal and written instructions.
3. Male or female subject between 18 to 50 years of age (inclusive) at the time of consent.
4. Subject's body mass index (BMI) must be at least 19.5 kg/m2 but no more than 37 kg/m2.
5. Female subject must have a negative serum pregnancy test at screening.
6. Female subjects of childbearing potential1 must agree to avoid pregnancy and use acceptable methods of birth control (see Section 24) from at least 60 days prior to screening and for at least 90 days after the last study drug administration.
7. Male subjects with female partner(s) of childbearing potential5 must agree to avoid fathering a child and use acceptable methods of birth control (see Section 24) from screening until at least 90 days after the last study drug administration.
8. Subject must meet the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition; Text Revision (DSM-IV-TR) criteria for a primary diagnosis of schizophrenia with the following subtypes: disorganized (295.10), catatonic type (295.20), paranoid (295.30), residual (295.60), or undifferentiated (295.90); and in the opinion of the Investigator has been clinically stable for the past 6 months.
9. Subject must have a Clinical Global Impression-Severity of Illness (CGI-S) score ≤ 4 (normal to moderately ill) at screening.
10. Subject must have a Positive and Negative Syndrome Scale (PANSS) total score ≤ 80 at screening.
11. Subject must have a score of ≤ 4 (normal to moderate) on the following PANSS items at screening:

    * P7 (hostility)
    * G8 (uncooperativeness)
12. Subject must be able and agree to remain off prior antipsychotic medication from clinic admission through Day 4.
13. Subject must have normal to mild symptoms on all individual items of the MSAS (< 2) and AIMS (< 3), and the clinical global assessment item of the BARS (< 3).
14. Subject is, in the opinion of the Investigator, generally healthy based on screening medical history, physical examination, neurological examination, vital signs, clinical laboratory values (hematology, serum chemistry, urinalysis, lipid panel, coagulation panel, and thyroid panel), and a 12-lead ECG.
15. Subject must be willing to stay within the clinic for the required period and return for follow-up visits.
16. Subject must possess an educational level and degree of understanding of English that enables them to communicate suitably with the Investigator and study coordinator.
17. Subject must agree to comply with all restrictions for the required length of time (see Section 10.5).

Exclusion Criteria:

1. Subject does not tolerate venipuncture or has poor venous access that would cause difficulty for collecting blood samples.
2. Subject has participated in an investigational drug study and received investigational drug within 30 days (or longer if the half-life is known to be ≥ 150 hours) prior to the screening visit, or who is currently participating in another clinical study. Subject has previously received study drug.
3. Subject has any clinically significant unstable medical condition or any clinically significant chronic disease that in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in the study:

   * a. Hematological (including deep vein thrombosis) or bleeding disorder, renal, metabolic, endocrine, pulmonary, gastrointestinal, urological, cardiovascular, hepatic, neurologic, or allergic disease (except for untreated, asymptomatic, seasonal allergies at time of dosing).
   * b. History of cancer or significant neoplasm.
   * c. Disorder or history of a condition, or previous gastrointestinal surgery (eg, cholecystectomy, vagotomy, bowel resection, or any surgical procedure) that may interfere with drug absorption, distribution, metabolism, excretion, gastrointestinal motility, or pH, or a clinically significant abnormality of the hepatic or renal system, or a history of malabsorption.
   * d. Known or suspected excessive alcohol consumption exceeding 14 drinks/week (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of the screening visit or a positive breath alcohol test at screening.
   * e. Subject has a clinically significant abnormal 12-lead ECG that may jeopardize the subject's ability to complete the study or a screening 12-lead ECG demonstrating any one of the following: heart rate > 100 beats per minute, QRS > 120 ms, QT interval corrected for heart rate using Fridericia's formula (QTcF) > 450 ms (males), QTcF > 470 ms (females), or PR > 220 ms.
4. Female subject who is pregnant or lactating.
5. Subject has a presence or history of a medically diagnosed, clinically significant psychiatric disorder (including mental retardation, schizoaffective disorder, schizophreniform disorder, psychotic depression, and bipolar disorder) other than schizophrenia.
6. Subject experienced an acute exacerbation of psychosis within the last 3 months or experienced an acute exacerbation of psychosis requiring hospitalization within the last 6 months.
7. Subject experienced an acute exacerbation of psychosis requiring change in antipsychotic medication (with reference to drug or dose) within the last 3 months.
8. Subject has a diagnosis or history of substance dependence (except nicotine ≤ 1 pack/day) or substance abuse (except cannabis) according to DSM IV-TR criteria ≤ 3 months prior to screening or a positive urine drug screen (except benzodiazepines) at screening.
9. Subject is at significant risk of harming himself or others according to the Investigator's judgment.
10. Subject has had past episodes of significant extrapyramidal symptoms (EPS) under current medication that required dose modification or the addition of anti-Parkinson's treatment within the last 6 months.
11. Subject is currently or has within 1 year before entering the study been treated with a depot antipsychotic medication.
12. Subject is under forced treatment.
13. Subject is taking aripiprazole at screening. Subject takes or has taken other disallowed recent or concomitant medications (see Section 10.5). Subjects must taper off schizophrenia medications by Day -1.
14. Subject has a history of allergic reaction to any medication or has a known or suspected sensitivity to any substance that is contained in the formulation.
15. Subject has any clinically significant abnormal laboratory values (hematology, serum chemistry, urinalysis, lipid panel, coagulation panel, and thyroid panel) (Note: clinically significant abnormal findings to be discussed with the Medical Monitor prior to including subject).
16. Subject has a history of hospitalization within 45 days prior to the screening visit.
17. Subject has a positive test for Hepatitis B surface antigen or Hepatitis C antibody at screening.
18. Subject has a positive test for Human Immunodeficiency Virus Type 1 or 2 (HIV-1 or HIV-2) at screening, or subject is known to have tested positive for Human Immunodeficiency Virus (HIV).
19. Subject has abnormal hepatic function tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT], bilirubin) or renal function (estimated creatinine clearance [CrCl] < 95 mL/min for males and < 85 mL/min for females based on serum creatinine using Modification of Diet in Renal Disease [MDRD]-glomerular filtration rate [GFR] method) at screening.
20. Subject has experienced significant blood loss (≥ 473 mL) or donated blood within 60 days prior to first dose of study drug; has donated plasma within 72 hours prior to the first dose of study drug or intends to donate plasma or blood or undergo elective surgery during study participation or within 60 days after the last study visit.
21. Subject consumes more than 300 mg of caffeine per day (5 cups of coffee or equivalent in caffeinated beverages).
22. Subject has used prescription or nonprescription drugs, vitamins, or dietary or herbal supplements within 14 days prior to dosing or anticipates the need for any medication during their participation in this study [exception: female subjects who are taking oral, patch, or intrauterine device (IUD) hormonal contraceptives, or progestin implant or injection]. Enzyme modulating herbal supplements (eg, Metabolife™) must be discontinued 30 days prior to the first dose of study drug.
23. Subject is a staff member or the relative of a staff member.
24. Subject is in the opinion of the Investigator, unsuitable in any other way to participate in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs), serious adverse events (SAEs), and AEs resulting in study discontinuation. | Up to 50 days
Absolute values and changes from baseline in clinical laboratory tests, vital signs, 12-lead electrocardiograms, and findings from neurological examinations. | Up to 50 days
  Absolute values and changes from baseline in clinical laboratory tests (hematology, serum chemistry, urinalysis, lipid panel, coagulation panel, and thyroid panel), vital signs (blood pressure [supine and standing], heart rate [supine and standing], respiration rate, and body temperature), 12-lead electrocardiograms (ECGs), and findings from neurological examinations.
Frequency of subjects with suicidal ideation or suicidal behavior using the Columbia-Suicide Severity Rating Scale (C-SSRS). | Up to 50 days

SECONDARY OUTCOMES:
Plasma SEP-363856 maximum observed concentration, area under the concentration-time curve, AUC0-inf, time of occurrence of Cmax, terminal elimination half-life, apparent clearance, and apparent volume of distribution. | Up to 50 days
  Plasma SEP-363856 maximum observed concentration (Cmax), area under the concentration-time curve (AUC0- last), AUC0-inf, time of occurrence of Cmax (tmax), terminal elimination half-life (t1/2), apparent clearance (CL/F), and apparent volume of distribution (Vz/F) following single oral dose administration of SEP-363856.
Plasma metabolite SEP-363854 Cmax, AUC0-last, AUC0-inf, tmax, and t1/2 following single oral dose administration of SEP-363856. | Up to 50 days
  Plasma metabolite SEP-363854 Cmax, AUC0-last, AUC0-inf, tmax, and t1/2 following single oral dose administration of SEP-363856.
Plasma metabolite to parent ratio for Cmax (MRCmax) and AUC0-inf (MRAUC0-inf) following single oral dose administration of SEP-363856. | Up to 50 days
  Plasma metabolite to parent ratio for Cmax (MRCmax) and AUC0-inf (MRAUC0-inf) following single oral dose administration of SEP-363856.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - California Clinical Trials Medical Group, Glendale, California
  - Collaborative Neuroscience Network, LLC, Long Beach, California

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com